CLINICAL TRIAL: NCT00131573
Title: Battery Powered Bion Clinical Investigation: Bion - An Implantable Microstimulator for the Chronic Treatment of Refractory Urinary Urgency-Frequency Syndrome
Brief Title: An Implantable Microstimulator for the Chronic Treatment of Urinary Urgency-Frequency Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-B-002
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Overactive Bladder
Keywords: Urgency-Frequency; Syndrome; Urinary; Refractory; Stimulation; Nerve; Neuromodulation; Microstimulator; bion; Pudendal; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stimulation On from Initial Activation up to the 12 month post-activation. Stimulation Off from 12 months post-activation until 45 days after the 12 month visit. Stimulation On from 45 days post 12 month visit and on.
  Interventions: Device: bion
- 2 (Sham Comparator): No stimulation until 45 days post-implant. Stimulation On from 45 days post-implant and on.
  Interventions: Device: bion

INTERVENTIONS:
Device: bion — battery powered bion microstimulator

SUMMARY:
The goal of this study is to investigate the safety and effectiveness of a new implanted device designed to treat Urinary Urgency-Frequency Syndrome.

ELIGIBILITY:
Key Inclusion criteria:

* Age 18 years and above.
* Diagnosed with urinary urgency-frequency syndrome.
* Have no reported history of urethral obstruction/stricture, bladder calculi or bladder tumor.
* Have normal upper urinary tract function.
* Be capable of giving informed consent.
* Be capable and willing to follow all study related procedures.

Key Exclusion Criteria:

* Have any active implantable device regardless of whether stimulation status is ON or OFF.
* Are pregnant as confirmed by a urine pregnancy test or plan to become pregnant during the following 12 month period.
* Less than one year post partum and/or are breast-feeding.
* Have any large passive implant that contains metal located within 30 cm of the chair pad while seated (e.g., hip replacement).
* Have conditions requiring magnetic resonance imaging (MRI) evaluation.
* Have conditions requiring diathermy procedures.
* Have an inability to operate the bion Remote Control and bion Recharging System either by self or caregiver.
* Have diabetes with peripheral nerve involvement or have severe uncontrolled diabetes.
* Have history of coagulopathy or bleeding disorder.
* Have pelvic pain in the absence of voiding dysfunction.
* Have anatomical restrictions such that the study device placement is not possible.
* Are currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function.
* Cannot independently comprehend and complete the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Baynham, PhD, Study Director — Boston Scientific, Neuromodulation
Locations (11):
- United States (11):
  - Arizona Health Sciences Center, Tucson, Arizona
  - The Department of Urology, Stanford University Medical Center, Stanford, California
  - Milestone Medical Research, Englewood, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cornerstone Medical Specialty Center, Woodbury, Minnesota
  - New York University, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Pelvic and Sexual Health Institute, Philadelphia, Pennsylvania
  - Dallas Center for Pelvic Medicine, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although enrollment numbers totaled 118 subjects, the total number of implanted subjects were used for the analysis. Total number of implanted subjects is 85.
Groups:
- Control: No stimulation until 45 days post-implant. Stimulation On from 45 days post-implant and on.
- Treatment: Stimulation On from Initial Activation up to the 12 month post-activation. Stimulation Off from 12 months post-activation until 45 days after the 12 month visit.
  Stimulation On from 45 days post 12 month visit and on.
Period: Overall Study
Arm/Group | Control | Treatment
Started | 46 | 39
Completed | 13 | 13
Not Completed | 33 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 46 | 39 | 85
Age, Customized [Mean (Standard Deviation); unit: Years] | 47.96 (11.66) | 46.64 (15.55) | 47.35 (13.53)
Sex/Gender, Customized [Number; unit: participants]
  Female | 39 | 33 | 72
  Male | 6 | 6 | 12
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Voids Per Day
Time Frame: 12 months
Measure: Median (Standard Deviation); unit: Average Number of Voids
Arm/Group | Treatment | Control
Number analyzed (Participants) | 39 | 46
Average Number of Voids | NA (NA) — This study was limited by poor adherence to the clinical protocol and by incomplete data recovery. Analysis of efficacy-related endpoints was not possible. | NA (NA) — This study was limited by poor adherence to the clinical protocol and by incomplete data recovery. Analysis of efficacy-related endpoints was not possible.

2. Primary Outcome: Freedom From Major Complications
Time Frame: 5 years
Measure: Number; unit: Number of Adverse Events
Arm/Group | Treatment | Control
Number analyzed (Participants) | 39 | 46
Number of Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Control | Treatment
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/39
Other Adverse Events (participants affected / at risk) | 30/46 | 21/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=46) | Treatment (N=39)
Defaecation Urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 2 (3)
Pelvi Floor Dyssynergia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adhesion (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Implant Site Haematoma (General disorders) | 0 (0) | 1 (1)
Implant site Pain (General disorders) | 4 (4) | 2 (3)
Implant site Swelling (General disorders) | 0 (0) | 2 (2)
No therapeutic response (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Therapeutic Product Ineffective (General disorders) | 10 (10) | 5 (5)
Therapeutic Response Decreased (General disorders) | 6 (9) | 5 (6)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Incision Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (3)
Device Breakage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — One non-serious device related unanticipated event occurred in the entire UF study. The event was related to broken bion during explant. Another non-serious device-related event of broken bion during explant occurred. No clinical outcome occured.
Device electrical Finding (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Device failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device Migration (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
Inappropriate Device Stimulation of Tissue (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Muscle Contractions involuntary (Nervous system disorders) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurological Symptom (Nervous system disorders) | 0 (0) | 1 (1)
Bladder Discomfort (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder Pain (Renal and urinary disorders) | 1 (1) | 2 (2)
Cystitis Interstitial (Renal and urinary disorders) | 2 (2) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Perineal Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was limited by poor adherence to the clinical protocol and by incomplete data recovery. Analysis of efficacy-related endpoints was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No